CLINICAL TRIAL: NCT00162656
Title: Treatment of Mature B-cell Lymphoma/Leukaemia A SFOP LMB 96/CCG 5961/UKCCSG NHL 9600 Cooperative Study
Brief Title: Treatment of Mature B-cell Lymphoma/Leukaemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAB LMB96
Record Dates: First submitted 2005-09-07; First posted 2005-09-13 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: B-Cell Lymphoma
Keywords: B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Standard LMB B (Active Comparator)
  Interventions: Drug: LMB B
- LMB B without COPADM3 (Experimental)
  Interventions: Drug: without COPADM3
- LMB B with half cyclophosphamide (Experimental)
  Interventions: Drug: half cyclophosphamide
- LMB B without COPADM3 and with half cyclophosphamide (Experimental)
  Interventions: Drug: half cyclophosphamide; Drug: without COPADM3
- LMB C standard (Active Comparator)
  Interventions: Drug: LMB C
- LMB C with mini CYVE and without 3 maintenance courses (Experimental)
  Interventions: Drug: mini CYVE, without 3 maintenance courses

INTERVENTIONS:
Drug: half cyclophosphamide
  Arms: LMB B with half cyclophosphamide; LMB B without COPADM3 and with half cyclophosphamide
Drug: without COPADM3
  Arms: LMB B without COPADM3; LMB B without COPADM3 and with half cyclophosphamide
Drug: mini CYVE, without 3 maintenance courses
  Arms: LMB C with mini CYVE and without 3 maintenance courses
Drug: LMB B
  Arms: Standard LMB B
Drug: LMB C
  Arms: LMB C standard

SUMMARY:
This is an international trial conducted by three cooperative groups: SFOP (France, Belgium, Netherlands), CCG (USA, Canada, Australia), and UKCCSG (UK and Ireland). Children with mature B-cell lymphoma/leukaemia are stratified into three different risk groups (A, B, C) and receive treatment of progressive intensity. Randomized trials in the 2 biggest groups (B and C) test whether "reduced" therapy is equivalent to standard intensive therapy (LMB-89 B and C) in terms of event free survival. The reason for the modification is to reduce the long term toxicity which includes cardiotoxicity, impaired fertility and secondary malignancy. In group B, the modifications of treatment consists of a reduction of cyclophosphamide in COPADM2 and/or the elimination of COPADM3. In group C, the modification consists in a reduction of the doses in the CYVE courses and the elimination of the last 3 courses of maintenance treatment

DETAILED DESCRIPTION:
Group B: Randomized trial with factorial design. The 4 treatment arms are standard LMB89 therapy B, reduction of cyclophosphamide (CPM) in COPADM2, deletion of COPADM3, both reduction and deletion. Randomization occurs following COPADM1 and is stratified for national group, histology (large cell; small non cleaved cell) and stage (Murphy I orII; Murphy III+LDH<2N; Murphy III+LDH>2N or Murphy IV).

The primary analysis questions are whether reducing CPM dose in COPADM2 results in a smaller long-term EFS whether omitting COPADM3 results in a smaller long-term EFS

Group C: Randomized trial. The 2 treatment arms are standard LMB89 therapy C versus reduction of CYVE + deletion of the last 3 maintenance courses. Randomization occurs following COPADM2 and is stratified for national group, histology (large cell; small non cleaved cell) and CNS disease.

The primary analysis question is whether reducing CYVE and omitting the last 3 maintenance courses result in a smaller long-term EFS than standard LMB 89 treatment C

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed B lineage non-Hodgkin's lymphoma with Revised European American Lymphoma (REAL) II 9 (diffuse large cell lymphoma), 10 (Burkitt's lymphoma), or 11 (high grade B cell lymphoma, Burkitt's like) or bone marrow > 5% L3 blasts.
* Pre treatment imaging studies adequate to document Murphy disease stage
* Group B and C patients are eligible for randomization (Therapy stratification by group : Group A=completely resected stage I or completely resected abdominal stage II lesions, Group B= All cases not eligible for Group A or Group C, Group C= Any CNS involvement and/or bone marrow involvement ³ 25% blasts)
* Patients should be available for a minimum follow up of 36 months
* Informed consent prior to study entry

Exclusion Criteria:

* Anaplastic large cell Ki 1 positive lymphomas
* Previous chemotherapy.
* Congenital immunodeficiency
* Prior organ transplantation
* Previous malignancy of any type
* Known HIV positivity

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 848 (Actual)
Dates: Start 1996-05; Primary Completion 2004-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Event free survival | 3 years
  Event free survival (event = progressive disease or relapse or second malignancy or death from any cause)

SECONDARY OUTCOMES:
Survival | 3 years
long term toxicity | 10 years
  long term toxicity: cardiotoxicity, impaired fertility, secondary malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Patte, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Mitchell S Cairo, MD, Principal Investigator — Morgan Stanley Childrens Hospital of New York Presbyterian, Columbia University; Mary Gerrard, MD, Principal Investigator — Sheffield Children's Hospital
Locations (3):
- Morgan Stanley Childrens Hospital of New York Presbyterian, New York, New York, United States
- Institut Gustave Roussy, Villejuif, France
- Sheffield Children's Hospital, Sheffield, United Kingdom

REFERENCES:
- [Derived] Frazer JK, Li KJ, Galardy PJ, Perkins SL, Auperin A, Anderson JR, Pinkerton R, Buxton A, Gross TG, Michon J, Leverger G, Weinstein HJ, Harrison L, Shiramizu B, Barth MJ, Goldman SC, Patte C, Cairo MS. Excellent outcomes in children and adolescents with CNS+ Burkitt lymphoma or other mature B-NHL using only intrathecal and systemic chemoimmunotherapy: results from FAB/LMB96 and COG ANHL01P1. Br J Haematol. 2019 Apr;185(2):374-377. doi: 10.1111/bjh.15520. Epub 2018 Aug 16. No abstract available. PMID 30117142